CLINICAL TRIAL: NCT05352477
Title: Double-blind Randomized Controlled Clinical Trial for Evaluating the Effects of Balneotherapy With Acquabios Thermal Water in Knee Osteoarthritis
Brief Title: Balneotherapy With Acquabios Thermal Water in Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Mario Fontana, Prof, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Acquabios1
Record Dates: First submitted 2022-04-13; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Knee Osteoarthritis
Keywords: Balneotherapy; Thermal water; Osteoarthritis; Musculoskeletal disease
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Musculoskeletal Diseases | interventions — Balneology

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balneotherapy with thermal water (Experimental): Daily balneotherapy with Acquabios thermal water at 33°C for 20 minutes each, for a total of 12 applications carried out over a period of 2 weeks
  Interventions: Other: Balneotherapy with thermal water
- Balneotherapy with tap water (Placebo Comparator): Daily balneotherapy with tap water at 33°C for 20 minutes each, for a total of 12 applications carried out over a period of 2 weeks
  Interventions: Other: Balneotherapy with tap water

INTERVENTIONS:
Other: Balneotherapy with thermal water — Bath with Acquabios thermal water at 33°C, 20 minutes daily for a total of 12 days, 6 days a week (from Monday to Saturday, Sundays excluded)
  Other Names: Acquabios thermal water of Minerbio (BO), Italy
  Arms: Balneotherapy with thermal water
Other: Balneotherapy with tap water — Bath with tap water at 33°C, 20 minutes daily for a total of 12 days, 6 days a week (from Monday to Saturday, Sundays excluded)
  Other Names: Tap water supplied by Minerbio water network
  Arms: Balneotherapy with tap water

SUMMARY:
The aim of the study is the evaluation of the effect of balneotherapy with Acquabios bicarbonate-alkaline-sodium thermal water in ameliorating some signs and symptoms of knee osteoarthritis in human subjects suffering from this disease

DETAILED DESCRIPTION:
This double-blind randomized controlled clinical trial is aimed to evaluate whether the balneotherapy with Acquabios thermal water is effective in improving some signs and symptoms of gonarthrosis in subjects affected by this disease.

The evaluated outcomes will be the reduction of pain and muscle-joint stiffness, the improvement of the joint range, the improvement of the quality of life, strength in the lower limbs and tolerance to physical exercise, the quality of walking and function in specific daily activities compared to the control group. Appropriated and validated tests will be used to evaluate the achievement of these outcomes.

The evaluation will be carried out on all patients enrolled in the study at the beginning, after the first week of treatment, after the second week of treatment and at the end of the study period (90 days after the first day of treatment). All eligible patients will be evaluated at the time of selection for weight, height, blood pressure, heart rate. These parameters will be evaluated and recorded on a specific form both during the enrollment and during all the visits planned for the follow-up. Each visit will last approximately 30 minutes.

The adverse reactions known for the balneotherapy with thermal water are the temporary reduction or increase of blood pression, thermal crisis and thermal reaction.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of right knee osteoarthritis
* Presence of pain characteristic of osteoarthritis of the right knee joint for at least 3 months
* Absence of severe disability
* Consent to treatment and participation in the study

Exclusion Criteria:

* Bilateral knee osteoarthrosis or left knee osteoarthritis
* Not eligilble for thermal balneotherapy treatments
* Previous arthroprotesis
* Previous balneotherapy treatments in last six months
* One or more steroid treatments in last two months
* One or more chondroprotective treatments, including infiltration with hyaluronic acid and similar in last six months
* One or more physiotherapy treatments in last two months, with the exception of exercises carried out individually at home
* Treatment with non-steroidal anti-inflammatory drugs in the last week
* One or more surgery on the lower limbs
* One or more trauma to the knee joint in the last 12 months
* Knee joint instability and / or intra-articular effusion before or during study participation
* Presence of palpable Baker's cyst
* Severe psychiatric or neurological conditions
* Being affected by severe chronic diseases: cardiovascular, respiratory, hepatic, cerebral, renal, juvenile diabetes, complicated diabetes mellitus, phlebopathies, systemic blood diseases, neoplasms
* Ongoing rheumatic diseases
* Being pregnant or breastfeeding
* Being suffering from severe acute pathologies

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Change of knee pain as assessed by Visual Analogue Scale | At baseline (T0), after 1 weeks (T1), after 2 weeks (T2),and after 3 months (T3) from the beginning of the study
  Knee pain change measured by the use of Visual Analogue Scale (VAS). VAS scale consists of a straight line segment (100 mm) at the ends of which there are the indications "no pain" (0 mm) and "the strongest pain imaginable" (100 mm). The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health) orientated from the left (best, 0) to the right (worst, 100).
Change of knee joint stiffness as assessed by Western Ontario and McMaster Universities.(WOMAC) osteoarthritis index | At baseline (T0), after 1 weeks (T1), after 2 weeks (T2) and after 3 months (T3) from the beginning of the study
  Knee joint stiffness change assessed by Western Ontario and McMaster Universities.(WOMAC) osteoarthritis index, a self-administered questionnaire. WOMAC questionnaire consists of 24 items divided into 3 subscales characterizing the patient's state of health: pain, joint stiffness and functionality. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function.
Change of knee range of motion change as assessed by the use of a universal goniometer | At baseline (T0), after 1 weeks (T1), after 2 weeks (T2) and after 3 months (T3) from the beginning of the study
  Knee range of motion change measured by the use of a universal goniometer
Change of walking quality as assessed by the 6-meters Walking Test. | At baseline (T0), after 1 weeks (T1), after 2 weeks (T2) and after 3 months (T3) from the beginning of the study
  Walking quality assessed by the 6-meters Walking Test, that evaluates the functional ability of walking by measuring the time required to walk 6 meters at a brisk pace. Each participants will be timed from the moment their foot cross the start line to the moment their foot cross the stop line placed at 6 meters from starting line.
Change of walking quality as assessed by Western Ontario and McMaster Universities (WOMAC) osteoarthritis score. | At baseline (T0), after 1 weeks (T1), after 2 weeks (T2) and after 3 months (T3) from the beginning of the study
  Change of walking quality assessed by Western Ontario and McMaster Universities (WOMAC) osteoarthritis score. WOMAC questionnaire consists of 24 items divided into 3 subscales characterizing the patient's state of health: pain, joint stiffness and functionality. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function.

SECONDARY OUTCOMES:
Change of quality of life as assessed by 36-Item Short Form Survey (SF-36) questionnaire | At baseline (T0) and after 3 months (T3) from the beginning of the study
  Quality of life assessed using 36-Item Short Form Survey (SF-36) questionnaire. The 36-Item Short Form Survey (SF-36) is a self-reported measure of health. It comprises 36 questions which cover eight domains of health: 1) Limitations in physical activities because of health problems; 2) Limitations in social activities because of physical or emotional problems; 3) Limitations in usual role activities because of physical health problems; 4) Bodily pain; 5) General mental health (psychological distress and well-being); 6) Limitations in usual role activities because of emotional problems; 7) Vitality (energy and fatigue); 8) General health perceptions. Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.
Change of lower limbs strength as assessed by 30-seconds Chair Stand Test (30-s CST) | At baseline (T0), after 1 weeks (T1), after 2 weeks (T2) and after 3 months (T3) from the beginning of the study
  Lower limbs strength assessed using 30-seconds Chair Stand Test (30-s CST), a performance based test. The 30-s CST is administered using a folding chair without arms, with seat height of 43.2 cm. The chair, with rubber tips on the legs, is placed against a wall to prevent it from moving. The 30-s CST involves recording the number of stands a person can complete in 30 seconds rather then the amount of time it takes to complete a pre-determined number of repetitions. That way, it is possible to assess a wide variety of ability levels with scores ranging from 0 for those who can not complete 1 stand to as many times as possible in 30 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Fontana, MD, Principal Investigator — University of Roma La Sapienza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomised trials. Trials. 2010 Mar 24;11:32. doi: 10.1186/1745-6215-11-32. PMID 20334632
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Cheleschi S, Gallo I, Tenti S. A comprehensive analysis to understand the mechanism of action of balneotherapy: why, how, and where they can be used? Evidence from in vitro studies performed on human and animal samples. Int J Biometeorol. 2020 Jul;64(7):1247-1261. doi: 10.1007/s00484-020-01890-4. Epub 2020 Mar 21. PMID 32200439
- [Background] D'Angelo D, Coclite D, Napoletano A, Fauci AJ, Latina R, Gianola S, Castellini G, Salomone K, Gambalunga F, Sperati F, Iacorossi L, Iannone P. The efficacy of balneotherapy, mud therapy and spa therapy in patients with osteoarthritis: an overview of reviews. Int J Biometeorol. 2021 Jul;65(7):1255-1271. doi: 10.1007/s00484-021-02102-3. Epub 2021 Mar 19. PMID 33740137